CLINICAL TRIAL: NCT06771973
Title: A Prospective Cohort Study Analysing Prediction of Successful Arteriovenous Fistula (AVF) Maturation Post Balloon Assisted Fistuloplasty With Duplex Ultrasound and Inflammatory Biomarkers
Brief Title: Ultrasound Prediction of Successful Balloon Assisted AVF Maturation
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24/YH/0247
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: End Stage Renal Disease (ESRD); Chronic Kidney Disease Requiring Hemodialysis
Keywords: arteriovenous fistula; AVF; CKD; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immature AVF (requiring BAM): Cohort to undergo BAM procedure. No additional interventions required.

SUMMARY:
An arteriovenous fistula (AVF) is created to allow for cleaning of the blood in patients with severe kidney disease. An artery and a vein are surgically connected, typically in the arm. This connection changes how the blood flows through the vessels, creating much higher flow in the arm vein than before the operation. Higher blood flow enables blood flow to be cleaned externally with a machine replacing the function of the kidneys. This process is known as dialysis. However, a period known as maturation is required before an AVF can be used in this way. During this time, the vessels grow in size and blood flow continues to increase. In some cases this does not happen and a procedure is required to help the AVF to mature.

AVFs not likely to mature may undergo a procedure, known as balloon assisted maturation (BAM), in which a balloon on the end of a catheter is inserted into the AVF vein and inflated. This is typically needed if an AVF is not likely to develop in a way that can be used for dialysis. Blood cleaning, or haemodialysis, is vital in patients with end stage renal disease, or kidney failure. Blood flow measurement using ultrasound, and routine blood test results, may help us predict which AVFs will respond better to BAM. Ultrasound can be used in the clinic setting and can provide the consultants responsible for the patients ongoing management with information that can enable decisions to be made at an early opportunity, and allowing the participants to be involved in future management decisions. This study aims to identify features of the blood flow following the BAM procedure that might be used to predict if the AVF will successfully mature.

DETAILED DESCRIPTION:
The study will be a prospective, longitudinal cohort study assessing maturation success following BAM procedures in immature AVFs. The primary outcome measure is successful AVF maturation at time of routine clinic appointment at 6 weeks post BAM procedure. Successful maturation is defined using a hybrid radiographic and clinical approach, namely a volume flow rate of ≥600ml/min, fistula vein diameter of ≥6mm combined with suitability for haemodialysis use as determined by clinician review. Failure to meet either criteria will be defined as failure to mature.

The primary objectives of the study will be met by comparing preoperative, postoperative and 6 week DUS values with maturation outcome. By comparing values obtained at these timepoints the investigators aim to identify factors predictive of maturation failure post BAM procedure. Neutrophil, platelet and lymphocyte values will be obtained from routine blood tests preoperatively and 2 week (+/- 1 week), and used to calculate both the neutrophil-lymphocyte (NLR) and platelet-lymphocyte ratios (PLR). Both ratios provide an indication of inflammatory status and will be compared with successful maturation post BAM procedure.

DUS scans will be performed pre- and post-BAM procedure in interventional radiology. Follow-up DUS scan will be performed when the participant is attending their 6 week routine clinical follow-up outpatient appointment. All scans will be performed by highly experienced clinical scientists using a single Philips Epiq 7 DUS scanner and L12-3 linear array transducer in accordance with a specified study scan protocol. A study preset will be used to standardise ultrasound settings. The DUS scan protocol will assess arterial inflow, arterio-venous anastomosis and venous outflow. Scan protocol and required measurements is the same for all DUS scans performed.

Arterial Inflow Peak systolic velocity (PSV), end diastolic velocity (EDV) and time averaged mean velocity (TAMV) will be measured in the brachial artery at each scan timepoint. TAMV will be measured across three cardiac cycles and combined with internal luminal diameter to calculate volume flow rate (Qa). Three measurements will be taken 10cm cranial to the antecubital fossa with a mean calculated. Sample volume gate for PSV measurements will be standardised at 1mm. Sample volume gate will be expanded to encompass the full vessel lumen for TAMV. TAMV sample volume gate will be recorded and remain consistent for subsequent scans for the same participant. Resistive (RI) and pulsatility indices (PI) will be calculated from the PSV and EDV values. All DUS-derived measurements will be recorded as absolute values and percentage change across DUS scans.

Access Anastomosis Anatomical location of the artery-vein anastomotic site will be recorded. PSV and EDV will be measured 5cm proximal to the anastomosis. Juxta-anastomotic PSV and EDV will also be measured. Stenoses present at the anastomosis will be graded using a ratio between PSV in the stenotic segment and the reference value 5cm proximally. Severity of stenoses will be recorded as a percentage. Minimal lumen diameter (MLD), defined as the narrowest luminal segment at the anastomosis will be recorded. Diameter of the arterial segment 2cm cranial to the anastomosis will be compared with the MLD to calculate the artery/fistula vein diameter ratio (A/V ratio).

Venous Outflow Venous outflow diameter and TAMV will be measured 10cm cranial to the arterial anastomosis, with venous Qa measured in the same way as for the brachial artery. Stenotic venous segments will be graded in the same way as the arterial inflow. Treatment of lesions as part of the BAM procedure will be noted from operative notes, and the treated lesions subsequently assessed. Residual stenosis, the presence of intimal hyperplasia and vein diameter will be measured at treatment site.

Neutrophil, lymphocyte and plasma values will be obtained from routine full blood count (FBC) results in the patient's electronic records. Neutrophil, lymphocyte and plasma values will be used to calculate neutrophil-to-lymphocyte (NLR) and plasma-to-lymphocyte ratios (PLR). Blood tests will be performed in accordance with standard of care. Patient age, sex, relevant medical history, current medication, and AVF configuration will be obtained from electronic patient records.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age) referred for BAM procedure due to immature native AVF
* AVFs with radio-cephalic or brachio-cephalic configuration
* AVF suitable for endovascular BAM procedure
* Patient is able to provide informed consent
* Patient is willing and able to comply with the study-related procedures

Exclusion Criteria:

* Brachio-basilic AVFs requiring transposition and superficialisation procedures during maturation phase
* Patients with arterio-venous grafts (AVGs) for vascular access
* Previous BAM procedures performed to facilitate maturation
* AVF unsuitable for BAM procedure or BAM procedure not performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with ESRD with immature AVFs requiring balloon assisted maturation procedures will be recruited from renal access clinics in a hospital setting
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-13 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Successful AVF maturation at time of routine clinic appointment at 6 weeks post BAM procedure | 6 weeks post BAM
  Hybrid radiographic and clinical approach, namely a volume flow rate of ≥600ml/min, fistula vein diameter of ≥6mm combined with suitability for haemodialysis use as determined by clinician review. Failure to meet either criteria will be defined as failure to mature.

IPD SHARING:
Plan to Share IPD: No